CLINICAL TRIAL: NCT00775203
Title: A Randomized, Double-blind, Two-arm Study Comparing the Efficacy and Safety of Trazodone Contramid® OAD and Placebo in the Treatment of Unipolar Major Depressive Disorder.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Labopharm Inc. (Industry)
Responsible Party: Vice-President Regulatory Affairs, Labopharm Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 04ACL3-001
Record Dates: First submitted 2008-10-17; First posted 2008-10-20 (Estimated); Results first posted 2010-04-07 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Major Depressive Disorder
Keywords: Unipolar
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Trazodone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Trazodone Contramid Once A Day (OAD) (Experimental)
  Interventions: Drug: Trazodone Hydrochloride (HCl) Extended-Release Tablets
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Trazodone Hydrochloride (HCl) Extended-Release Tablets
  Other Names: Oleptro
  Arms: Trazodone Contramid Once A Day (OAD)
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study was to demonstrate efficacy, safety and clinical benefit of Trazodone Contramid® OAD (Once A Day) in the treatment of Unipolar Major Depressive Disorder (MDD).

DETAILED DESCRIPTION:
This two-arm, multicentre, randomized, placebo-controlled, double-blind, parallel-design study consisted of a baseline phase (screening and wash-out) and a double-blind randomized phase (randomization to Trazodone Contramid® OAD or placebo). The total study duration including wash-out of prohibited medications was approximately 11 weeks; the total duration of the randomized phase was 8 weeks (titration: 2 weeks + treatment: 6 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Males or females.
* Aged 18 years or older.
* Fulfills Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV) criteria for Unipolar Major Depressive Disorder (MDD) (Axis I) as confirmed by the Mini-International Neuropsychiatric Interview (MINI).
* The primary DSM-IV Axis I diagnosis should be MDD (296.22, 296.23, 296.32, 296.33); any subject meeting criteria for another, non excluded Axis I disorder, must demonstrate MDD as the primary disorder.
* The current episode of MDD should have lasted for a minimum of 1 month, whether the patient has been diagnosed with one single or recurrent episodes.
* Presence of dysphoria for most days over the past four weeks.
* Montgomery-Åsberg Depression Rating Scale (MADRS) total score of at least 26 at screening and baseline.
* Oral and written language comprehension at a level sufficient to comply with the protocol and to complete study-related materials.
* Sign and date a written Informed Consent Form (ICF) approved by a Research Ethic Board (REB) which has also been signed and dated by the Investigator prior to study participation.

Exclusion Criteria:

* DSM-IV Major Depressive Disorder Specifiers: [a] With Catatonic Features; [b] With Postpartum Onset; [c] With Seasonal Pattern;
* Presence of any of the following DSM-IV Axis I disorders: generalized anxiety disorder, panic disorder, social phobia, obsessive-compulsive disorder, post-traumatic stress disorder, eating disorder, bipolar disorder, alcohol/substance abuse or dependence (caffeine and nicotine allowed), any psychotic disorder.
* Depression secondary to stroke, cancer or other severe medical illnesses.
* Positive urine drug screen at screening visit.
* History or present condition of any DSM-IV Axis II disorder.
* History of treatment refractory major depressive episodes defined as incomplete or no therapeutic response to two prior courses of at least one month of conventional antidepressant drug treatment in adequate dosages.
* Currently in psychotherapy (at least one session in the past month with a plan for continuing) with a licensed/registered/certified mental health provider, marriage counselor, or family therapist.
* Meet criteria for high suicide risk on the MINI suicide scale, or in the opinion of the investigator is inappropriate for the trial due to clinically significant suicidal or homicidal potential.
* Require hospitalization for treatment of the current episode of depression.
* Uncorrected hypo- or hyperthyroidism.
* A history of seizures other than pediatric febrile seizure.
* A history of cardiac arrythmias requiring therapy.
* A history of myocardial infarction within 1 year before screening.
* Clinically significant abnormal findings of Electrocardiography (ECG), laboratory parameters.
* Unwilling to discontinue use of any antidepressants, including herbal remedies, for a minimum of 5 drug half-lives prior to screening.
* Unwilling to discontinue use of prohibited medications for a minimum of 5 drug half-lives prior to screening.
* Treatment within the last 3 weeks with Monoamine Oxidase (MAO) inhibitors.
* Use of the following concomitant treatment during the study:

  * medications causing QT prolongation (e.g. amiodarone, droperidol, erythromycin).
  * medications causing PR prolongation (e.g. digoxin).
  * Anti -psychotics (e.g. haloperidol).
  * protease inhibitors such as ritonavir and indinavir.
* Hormonal treatment (e.g. estrogen, oral contraceptives) which has started within 3 months of study entry.
* Treatment with another investigational agent within the last 30 days.
* Known and documented allergy to trazodone or any structurally similar drugs.
* Previous failure of treatment with trazodone, or previous discontinuation of treatment with trazodone due to Adverse Events.
* Bowel disease causing malabsorption.
* Serious, unstable illnesses during the 3 months before screening including but not limited to: hepatic, renal, gastroenterologic, respiratory, cardiovascular (including ischemic heart disease), endocrinologic, neurologic, immunologic or hematological disease.
* Pregnant or lactating, or is of childbearing potential and not willing to use an approved method of contraception.
* Significant liver disease, defined as active hepatitis or elevated liver enzymes >3 times the upper boundary of the normal range.
* Significant renal disease, defined as Blood Urea Nitrogen (BUN) and/or creatinine >3 times the upper boundary of the normal range clearance.
* Any other condition that, in the opinion of the investigators, would adversely affect the patient's ability to complete the study or its measures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 412 (Actual)
Dates: Start 2007-06; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (36):
- United States (28):
  - Birmingham, Alabama
  - Mesa, Arizona
  - Beverly Hills, California
  - Burbank, California
  - San Diego, California
  - Denver, Colorado
  - Gainesville, Florida
  - Hialeah, Florida
  - Jacksonville, Florida
  - Orlando, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Marietta, Georgia
  - Smyrna, Georgia
  - Libertyville, Illinois
  - Indianapolis, Indiana
  - Overland Park, Kansas
  - Clementon, New Jersey
  - Brooklyn, New York
  - New York, New York
  - Beachwood, Ohio
  - Cincinnati, Ohio
  - Dayton, Ohio
  - Oklahoma City, Oklahoma
  - Philadelphia, Pennsylvania
  - Bellaire, Texas
  - San Antonio, Texas
  - Woodstock, Vermont
- Canada (8):
  - Kelowna, British Columbia
  - Penticton, British Columbia
  - Mount Pearl, Newfoundland and Labrador
  - Hamilton, Ontario
  - Oakville, Ontario
  - Gatineau, Quebec
  - Saint-Léonard, Quebec
  - Sherbrooke, Quebec

REFERENCES:
- [Result] Sheehan DV, Croft HA, Gossen ER, Levitt RJ, Brulle C, Bouchard S, Rozova A. Extended-release Trazodone in Major Depressive Disorder: A Randomized, Double-blind, Placebo-controlled Study. Psychiatry (Edgmont). 2009 May;6(5):20-33. PMID 19724732
- See also: Approved labelling — http://dailymed.nlm.nih.gov/dailymed/drugInfo.cfm?id=15386

RESULTS

PARTICIPANT FLOW:
Groups:
- Trazodone Contramid OAD: Subjects with Major Depressive Disorder who were randomized to Trazodone Contramid OAD. Dose was titrated to each subject optimal dose every 3 to 4 days by 75 mg increments from a starting dose of 150 mg to a maximum daily dose of 375 mg. At each dosing step, if a dose was not well tolerated after 2 days, subjects had the option to decrease to the previous dose. Patients then continued six weeks of treatment; further dose adjustments were allowed based on efficacy and tolerability.
- Placebo: Subjects with Major Depressive Disorder who were randomized to Placebo to match Trazodone Contramid OAD.
Period: Overall Study
Arm/Group | Trazodone Contramid OAD | Placebo
Started | 206 | 206
Received Study Medication | 202 | 204
Completed | 144 | 163
Not Completed | 62 | 43
Not completed — Adverse Event | 25 | 6
Not completed — Lack of Efficacy | 8 | 9
Not completed — Withdrawal by Subject | 11 | 9
Not completed — Lost to Follow-up | 11 | 15
Not completed — Administrative reason | 2 | 0
Not completed — Noncompliance | 4 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Entered other study | 1 | 0
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Trazodone Contramid OAD | Placebo | Total
Number analyzed (Participants) | 202 | 204 | 406
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 2 | 2
  Between 18 and 65 years | 193 | 186 | 379
  >=65 years | 9 | 16 | 25
Age Continuous [Mean (Standard Deviation); unit: years] | 43.8 (12.83) | 44.0 (13.45) | 43.9 (13.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 129 | 131 | 260
  Male | 73 | 73 | 146
Region of Enrollment [Number; unit: participants]
  United States | 169 | 166 | 335
  Canada | 33 | 38 | 71

OUTCOME MEASURES:

1. Primary Outcome: Change in Hamilton Depression Scale (HAMD-17) Total Score From Baseline
Description: The Hamilton Depression Rating Scale 17 items [HAMD-17] is a 17-item scale that evaluates depressed mood, vegetative and cognitive symptoms of depression, and co-morbid anxiety symptoms. The 17 items are rated on either a 5-point (0-4) or a 3-point (0-2) scale. In general, the 5 point scale items use a rating of 0=absent; 1=doubtful to mild; 2=mild to moderate; 3=moderate to severe; 4=very severe. The 3-point scale items use a rating of 0=absent; 1=probable or mild; 2=definite. The total HAMD-17score ranges from 0 (not ill) to 52 (severely ill).
Time Frame: Baseline to Week 8
Population: Full analysis (intent-to-treat [ITT]) population is defined as all randomized patients who received any study medication and had a baseline and at least one post-baseline HAMD-17 assessment. Week 8 Last Observation Carried Forward (LOCF): Trazodone = 202, placebo = 204.
Measure: Mean (Standard Deviation); unit: Points on HAMD-17 scale
Arm/Group | Trazodone Contramid OAD | Placebo
Number analyzed (Participants) | 202 | 204
Points on HAMD-17 scale
  Baseline | 23.2 (4.16) | 22.4 (4.43)
  Week 8 or LOCF | 11.8 (7.99) | 13.2 (8.06)
  Change from baseline | -11.4 (8.20) | -9.3 (7.94)
Statistical Analysis 1: Comparison: Trazodone Contramid OAD vs Placebo; The primary null hypothesis for the HAMD-17 total score is that there is no difference between the Trazodone Contramid® OAD group and the placebo group at Week 8. A sample size of 133 in each group will have 90% power to detect a difference in the absolute mean Hamilton Rating Scale for Depression (HAMD-17) change from baseline of 3.0 units assuming that the common standard deviation is 7.5 using a two-group t-test with a 0.05 two-sided significance level; Test type: Superiority or Other; p = 0.0119, ANCOVA; ANCOVA with treatment and study center as categorical factors and HAMD-17 baseline as covariate

2. Secondary Outcome: HAMD-17 Responders at Each Visit
Description: Number of patients who show a response (defined as at least a 50% reduction from baseline in HAMD-17 score) at each post-baseline visit.
Time Frame: Weeks 1, 2, 3, 4, 6, 8
Population: Full analysis (intent-to-treat [ITT]) population is defined as all randomized patients who received any study medication and had a baseline and at least one post-baseline HAMD-17 assessment. Last Observation Carried Forward (LOCF).
Measure: Number; unit: Participants
Arm/Group | Trazodone Contramid OAD | Placebo
Number analyzed (Participants) | 202 | 204
Participants
  ≥50% reduction in HAMD-17 at Week 1 (n=197, n=199) | 25 | 19
  ≥50% reduction in HAMD-17 at Week 2 (n=201, n=203) | 63 | 41
  ≥50% reduction in HAMD-17 at Week 3 (n=202, n=204) | 89 | 53
  ≥50% reduction in HAMD-17 at Week 4 (n=202, n=204) | 95 | 74
  ≥50% reduction in HAMD-17 at Week 6 (n=202, n=204) | 100 | 81
  ≥50% reduction in HAMD-17 at Week 8 (n=202, n=204) | 109 | 84

3. Secondary Outcome: HAMD-17 Remitters at Each Visit
Description: Number of patients who are remitters (defined as patients who achieved a HAMD-17 total score ≤7) at each post-baseline visit.
Time Frame: Weeks 1, 2, 3, 4, 6, 8
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Trazodone Contramid OAD | Placebo
Number analyzed (Participants) | 202 | 204
Participants
  Number of remitters at Week 1 (n=197, n=199) | 10 | 9
  Number of remitters at Week 2 (n=201, n=203) | 29 | 24
  Number of remitters at Week 3 (n=202, n=204) | 51 | 32
  Number of remitters at Week 4 (n=202, n=204) | 61 | 43
  Number of remitters at Week 6 (n=202, n=204) | 66 | 47
  Number of remitters at Week 8 (n=202, n=204) | 72 | 65

4. Secondary Outcome: Change in HAMD-17 Depressed Mood Item (Item 1) Score From Baseline to Each Visit
Description: Change from baseline in the HAMD-17, item 1: Depressed Mood item, at each post-baseline visit. The Depressed Mood item is rated on a 5-point scale ranging from rating of 0=absent; to 4=very severe.
Time Frame: Baseline to Weeks 1, 2, 3, 4, 6, 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Points on the HAMD scale
Arm/Group | Trazodone Contramid OAD | Placebo
Number analyzed (Participants) | 202 | 204
Points on the HAMD scale
  Change in score at Week 1 (n=197, n=199) | -0.7 (0.89) | -0.5 (0.74)
  Change in score at Week 2 (n=201, n=203) | -1.1 (1.13) | -0.8 (0.95)
  Change in score at Week 3 (n=202, n=204) | -1.4 (1.18) | -1.0 (1.08)
  Change in score at Week 4 (n=202, n=204) | -1.5 (1.21) | -1.2 (1.12)
  Change in score at Week 6 (n=202, n=204) | -1.5 (1.18) | -1.3 (1.15)
  Change in score at Week 8 (n=202, n=204) | -1.6 (1.29) | -1.3 (1.22)

5. Secondary Outcome: Change in Montgomery-Åsberg Depression Rating Scale (MADRS) Total Score From Baseline
Description: The Montgomery-Åsberg Depression Rating Scale (MADRS) is a 10 item clinician-administered depression rating scale. The 10 items (apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts) are rated on a scale ranging from 0 (low severity/difficulty) to 6 (high severity/difficulty) with anchors at 2-point intervals. The overall total score range is from 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms).
Time Frame: Baseline to Week 8
Population: Full analysis (intent-to-treat [ITT]) population is defined as all randomized patients who received any study medication and had a baseline and at least one post-baseline HAMD-17 assessment. MADRS Week 8 Observed Cases: Trazodone = 178, placebo = 182.
Measure: Mean (Standard Deviation); unit: Units on MADRS scale
Arm/Group | Trazodone Contramid OAD | Placebo
Number analyzed (Participants) | 178 | 182
Units on MADRS scale
  Baseline (n=202, n=204) | 32.6 (4.07) | 31.9 (4.33)
  Week 8 (n=178, n=182) | 16.0 (11.24) | 17.7 (11.62)
  Change from baseline (n=178, n=182) | -16.6 (11.27) | -14.1 (11.27)

6. Secondary Outcome: Change From Baseline in Clinical Global Impression of Severity (CGI-S) to Each Visit
Description: The CGI-Severity (CGI-S) consists of one question for the investigator: "Considering your total clinical experience with this particular population, how mentally ill is the patient at this time?" which is rated on the following seven-point scale: 1=normal, not ill at all; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most extremely ill patients.
Time Frame: Baseline to Weeks 1, 2, 3, 4, 6, 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on CGI-S scale
Arm/Group | Trazodone Contramid OAD | Placebo
Number analyzed (Participants) | 202 | 204
Units on CGI-S scale
  Change in CGI-S score at Week 1 (n=197, n=199) | -0.6 (0.72) | -0.5 (0.75)
  Change in CGI-S score at Week 2 (n=201, n=203) | -1.0 (1.02) | -0.8 (0.98)
  Change in CGI-S score at Week 3 (n=202, n=204) | -1.4 (1.16) | -1.1 (1.12)
  Change in CGI-S score at Week 4 (n=202, n=204) | -1.6 (1.22) | -1.3 (1.17)
  Change in CGI-S score at Week 6 (n=202, n=204) | -1.7 (1.24) | -1.4 (1.24)
  Change in CGI-S score at Week 8 (n=202, n=204) | -1.7 (1.36) | -1.4 (1.37)

7. Secondary Outcome: Clinical Global Impression - Improvement of Illness (CGI-I) Score at Last Study Visit
Description: The CGI-Improvement of Illness (CGI-I) consists of one question for the investigator: "Compared to his condition at the start of the study, how much has this patient changed?" which is rated on the following seven-point scale 1=very much improved; 2=much improved; 3=minimally improved; 4=no change from baseline; 5=minimally worse; 6= much worse; 7=very much worse.
Time Frame: Week 8
Population: Full analysis (intent-to-treat [ITT]) population is defined as all randomized patients who received any study medication and had a baseline and at least one post-baseline HAMD-17 assessment. CGI-I Week 8 Observed Cases: Trazodone = 178, placebo = 182.
Measure: Mean (Standard Deviation); unit: Units on the CGI-I scale
Arm/Group | Trazodone Contramid OAD | Placebo
Number analyzed (Participants) | 178 | 182
Units on the CGI-I scale | 2.4 (1.23) | 2.5 (1.32)

8. Secondary Outcome: Patient Global Impression - Improvement of Illness (PGI-I) Score at Last Study Visit
Description: The PGI-Improvement of Illness (PGI-I) consists of one question for the patient: "Since the start of the study, my overall status with regard to depression is?" which is rated on the following seven-point scale 1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6= much worse; 7=very much worse.
Time Frame: Week 8
Population: Full analysis (intent-to-treat [ITT]) population is defined as all randomized patients who received any study medication and had a baseline and at least one post-baseline HAMD-17 assessment. PGI-I Week 8 Observed Cases: Trazodone = 176, placebo = 183.
Measure: Mean (Standard Deviation); unit: Units on PGI-I scale
Arm/Group | Trazodone Contramid OAD | Placebo
Number analyzed (Participants) | 176 | 183
Units on PGI-I scale | 2.6 (1.19) | 2.8 (1.35)

9. Secondary Outcome: Clinical Global Impression - Improvement of Illness (CGI-I) Responders at Last Study Visit
Description: Patients were responders if the CGI-I rating was "Much Improved" or "Very Much Improved". The CGI-Improvement of Illness (CGI-I) consists of one question for the investigator: "Compared to his condition at the start of the study, how much has this patient changed?" which is rated on the following seven-point scale 1=very much improved; 2=much improved; 3=minimally improved; 4=no change from baseline; 5=minimally worse; 6= much worse; 7=very much worse. Results are expressed in number of patients.
Time Frame: Week 8
Population: Full analysis (intent-to-treat [ITT]) population is defined as all randomized patients who received any study medication and had a baseline and at least one post-baseline HAMD-17 assessment. CGI-I Responders Week 8 Observed Cases: Trazodone = 180, placebo = 183.
Measure: Number; unit: participants
Arm/Group | Trazodone Contramid OAD | Placebo
Number analyzed (Participants) | 180 | 183
participants | 96 | 89

10. Secondary Outcome: Patient Global Impression - Improvement of Illness (PGI-I) Responders at Last Study Visit
Description: Patients were responders if the PGI-I rating was "Much Improved" or "Very Much Improved". The PGI-Improvement of Illness (PGI-I) consists of one question for the patient: "Since the start of the study, my overall status with regard to depression is?" which is rated on the following seven-point scale 1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6= much worse; 7=very much worse. Results are expressed in number of patients.
Time Frame: Week 8
Population: Full analysis (intent-to-treat [ITT]) population is defined as all randomized patients who received any study medication and had a baseline and at least one post-baseline HAMD-17 assessment. PGI-I Responders Week 8 Observed Cases: Trazodone = 176, placebo = 183.
Measure: Number; unit: participants
Arm/Group | Trazodone Contramid OAD | Placebo
Number analyzed (Participants) | 176 | 183
participants | 90 | 80

11. Secondary Outcome: Overall Quality of Sleep at Each Visit
Description: Overall Quality of Sleep was measured on a 4-point rating scale ranging from 1 = very poor to 4 = excellent in response to the question: "Since the last study visit, how would you rate the overall quality of your sleep?".
Time Frame: Weeks 1, 2, 3, 4, 6, 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | Trazodone Contramid OAD | Placebo
Number analyzed (Participants) | 202 | 204
Points on a scale
  Score at Baseline (n=202, n=204) | 1.6 (0.65) | 1.6 (0.70)
  Score at Week 1 (n=196, n=199) | 0.7 (0.90) | 0.4 (0.83)
  Score at Week 2 (n=200, n=203) | 0.8 (0.97) | 0.7 (0.99)
  Score at Week 3 (n=201, n=204) | 0.9 (1.00) | 0.7 (1.00)
  Score at Week 4 (n=201, n=204) | 1.0 (1.02) | 0.7 (1.02)
  Score at Week 6 (n=201, n=204) | 1.0 (1.01) | 0.9 (1.04)
  Score at Week 8 (n=201, n=204) | 1.0 (1.05) | 0.8 (1.10)

12. Secondary Outcome: Trouble Falling Asleep at Each Visit
Description: Trouble Falling Asleep was measured on a 4-point rating scale ranging from 1 = never to 4 = always in response to the question: "Since the last study visit, how often did you experience trouble falling asleep?".
Time Frame: Weeks 1, 2, 3, 4, 6, 8
Population: Full Analysis set (intent-to-treat [ITT]) population is defined as all randomized patients who received any study medication and had a baseline and at least one post-baseline HAMD-17 assessment. Last Observation Carried Forward (LOCF).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Trazodone Contramid OAD | Placebo
Number analyzed (Participants) | 202 | 204
Units on a scale
  Score at Baseline (n=202, n=204) | 3.0 (0.86) | 2.9 (0.91)
  Score at Week 1 (n=196, n=199) | 2.5 (1.02) | 2.6 (0.98)
  Score at Week 2 (n=200, n=203) | 2.3 (0.93) | 2.5 (0.96)
  Score at Week 3 (n=201, n=204) | 2.2 (0.90) | 2.3 (0.99)
  Score at Week 4 (n=201, n=204) | 2.1 (0.89) | 2.3 (0.95)
  Score at Week 6 (n=201, n=204) | 2.1 (0.89) | 2.3 (0.95)
  Score at Week 8 (n=201, n=204) | 2.1 (0.85) | 2.3 (0.95)

13. Secondary Outcome: Awakening During the Night at Each Visit
Description: Awakening during the night was measured on a 4-point rating scale ranging from 1 = never to 4 = always in response to the question: "Since the last study visit did you awaken during the night?".
Time Frame: Weeks 1, 2, 3, 4, 6, 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Trazodone Contramid OAD | Placebo
Number analyzed (Participants) | 202 | 204
Units on a scale
  Score at Baseline (n=202, n=204) | 3.2 (0.78) | 3.2 (0.78)
  Score at Week 1 (n=196, n=199) | 2.4 (0.96) | 2.7 (0.85)
  Score at Week 2 (n=200, n=203) | 2.4 (0.94) | 2.5 (0.92)
  Score at Week 3 (n=201, n=204) | 2.2 (0.91) | 2.6 (0.90)
  Score at Week 4 (n=201, n=204) | 2.2 (0.89) | 2.6 (0.93)
  Score at Week 6 (n=201, n=204) | 2.2 (0.94) | 2.5 (0.95)
  Score at Week 8 (n=201, n=204) | 2.2 (0.89) | 2.5 (0.95)

14. Secondary Outcome: Discontinuation Due to Lack of Efficacy
Description: Number of patients who discontinued due to lack of efficacy during the whole study period (8 weeks).
Time Frame: Baseline to Week 8
Population: Safety population is defined as all randomized patients who received any study medication.
Measure: Number; unit: participants
Arm/Group | Trazodone Contramid OAD | Placebo
Number analyzed (Participants) | 202 | 204
participants | 8 | 9

ADVERSE EVENTS:
Time Frame: 8 weeks (plus an additional 30 days for SAEs only)
Arm/Group | Trazodone Contramid OAD | Placebo
Serious Adverse Events (participants affected / at risk) | 4/202 | 2/204
Other Adverse Events (participants affected / at risk) | 168/202 | 122/204
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trazodone Contramid OAD (N=202) | Placebo (N=204)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Viral pericarditis (Infections and infestations) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trazodone Contramid OAD (N=202) | Placebo (N=204)
Vision blurred (Eye disorders) | 11 (12) | 0 (0)
Constipation (Gastrointestinal disorders) | 16 (17) | 4 (7)
Diarrhea (Gastrointestinal disorders) | 19 (23) | 23 (29)
Dry mouth (Gastrointestinal disorders) | 51 (58) | 26 (26)
Nausea (Gastrointestinal disorders) | 42 (51) | 26 (30)
Fatigue (General disorders) | 30 (34) | 17 (17)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (15) | 7 (8)
Dizziness (Nervous system disorders) | 50 (57) | 25 (25)
Headache (Nervous system disorders) | 67 (89) | 55 (98)
Sedation (Nervous system disorders) | 34 (39) | 7 (10)
Somnolence (Nervous system disorders) | 63 (80) | 32 (36)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to submitting results communications, the investigator shall allow Labopharm at least 60 days to review the proposed communication. If the proposed publication/disclosure risks Labopharm's ability to patent any invention related to the study, the publication or disclosure will be modified/delayed to allow Labopharm to seek patent protection. This statement does not give Labopharm any editorial rights other than to restrict the disclosure of Labopharm's confidential information.